CLINICAL TRIAL: NCT06609070
Title: CHG0521 Oral Coating; TSCC
Brief Title: CHG0521 Oral Coating in Patients with Solid Tissue Tumor/Recurrent/Metastatic TSCC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, jianwen guo, MD, Chief TCM physician, Guangzhou University of Traditional Chinese Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZF2024-260-01
Record Dates: First submitted 2024-09-20; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Squamous Cell Carcinoma; Squamous Cell Carcinoma of the Oral Cavity
MeSH Terms: conditions — Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Drug: CHG0521 Oral Coating (Experimental): LSCC subjects who are not suitable for surgery after evaluation, or have surgical indications, do not agree to surgical treatment, or patients with recurrence and metastasis after surgery no longer have surgery.
  Interventions: Drug: CHG0521 Oral Coating

INTERVENTIONS:
Drug: CHG0521 Oral Coating — The subjects will receive an oral coating of CHG0521 in the form of drops, in addition to the clinician's standard treatment regimen, for a duration of 6 months or until confirmed progression, unacceptable toxicity, or any criteria for withdrawal from the trial.

SUMMARY:
This is a prospective single-arm loading test study of CHG0521 oral coating in patients with solid tissue tumor/recurrent/metastatic TSCC

ELIGIBILITY:
Inclusion Criteria:

* 1. Age range: 18-80 years, encompassing both males and females. 2. Confirmation of tongue squamous cell carcinoma through histopathology or cytology is required.

  3. Patients who are deemed unsuitable for surgery, have surgical indications but decline the treatment, or experience relapse and metastasis after surgery with no further surgical options available.

  4. No concurrent use of other traditional Chinese medicine orally or externally within the past 3 months.

  5. Presence of at least one measurable lesion according to RECIST 1.1 criteria. 6. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.

  7. Expected survival time should be equal to or greater than 3 months. 8. Liver function indicators: total bilirubin level ≤1.5 times the upper limit of normal (ULN), AST and ALT levels ≤2.5 times ULN (or ≤5 times ULN in case of liver metastasis).

  9.Renal function indicators: serum creatinine (CRE) ≤1.5×ULN and calculated creatinine clearance (using Cockcroft-Gault formula) ≥60 ml/min.

  10.The functionality of vital organs should be essentially normal.

Exclusion Criteria:

* 1. Patients with tongue squamous cell carcinoma who have undergone tumor resection without any residual tumor; 2. Patients with a known allergy to any therapeutic ingredient or a history of hypersensitivity or allergic constitution; 3. Patients who have experienced a severe infection within 4 weeks prior to the first use of the investigational drug, and whose common adverse reaction criteria were graded as >2; 4. Patients with a history of immune deficiency, organ transplantation, or allogeneic bone marrow transplantation; 5. Patients currently enrolled in another concurrent clinical study; 6. Pregnant and lactating women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 24 weeks
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: at least 30% decrease in the sum of diameters of target lesions) per RECIST 1.1.

SECONDARY OUTCOMES:
QOL | 24 weeks
  Washington Quality of Life Score
PCR | 24 weeks
  Pathologic Complete Response
DRR | 24 weeks
  Disease Recurrence Rate
OS | 1 year
  Overall Survival
AEs | 1 year
  Incidence and severity of adverse events

IPD SHARING:
Plan to Share IPD: Undecided